CLINICAL TRIAL: NCT03361527
Title: Evaluation of a Binaural Beamformer (StereoZoom) in a Virtual Acoustic Environment and in Real Life
Status: Completed | Type: Observational
Sponsor: Advanced Bionics AG (Industry)
Responsible Party: Sponsor
Other Study IDs: ABERC-14-09-01
Record Dates: First submitted 2015-11-23; First posted 2017-12-05 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Sensory Hearing Loss
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: binaural beamformer — Each study participant will use an Advacned Bionics Naida CI Q90 loaner processor during the course of the study, an Advanced Bionics MyPilot remote control and- if applicable- a SmartPhone. the processors will be programmed with SoundWave and BEPSnet.

SUMMARY:
The goal of the study is to determine the benefit in speech intelligibility of the BBF and the MBF compared to an omni-directional microphone in different noise conditions. Secondary objective is to determine if there is a subjective preference for one of the microphone settings in different noise conditions.

DETAILED DESCRIPTION:
Study participants will be invited for two appointments. In the first appointment test will be performed inside the lab (lab measurements) and outside the lab (real life measurements) and in the second appointment test will be performed in the lab. In between appointments participants are asked to try the Naida CI Q90 at home and in their familiar surroundings for 2-4 weeks (home trial).

Lab measurements:

The Oldenburg Sentence Test will be used as speech signal to determine the speech reception threshold (SRT) for each background noise with an adaptive procedure. The overall level of the noise will be held constant while the level of the speech signal will be adapted depending on the words understood correctly for each sentence.

In addition to the objective speech intelligibility measurements the three microphone settings will also be assessed subjectively. For each background noise scenario the Oldenburg sentences will be presented successively from the frontal loudspeaker. The experimenter will switch between two programs on the participant's processor who then compares the two different microphone settings of these programs. Three paired comparisons will be performed: omni-directional vs. MBF, omni-directional vs. BBF and MBF vs. BBF. The comparisons will be made with regards to speech intelligibility, noise suppression and overall preference in each situation.

Real life measurements:

Even though the results obtained in the lab present a good approximation to real-life performance both beam former options should also be tested outside the lab and in everyday life. In a guided tour the experimenter will take the study participant to noisy places in Zürich, if possible to the same or similar places in which the lab recordings were made. The same paired comparisons as in the lab will be performed with the experimenter talking to the participant or reading a story aloud.

Home trial:

Finally, the study participant should evaluate all three microphone settings for 2-4 weeks during activities in their familiar surroundings, i.e. having a conversation with one or more persons at home, in the tram, in a restaurant, attending a meeting at work, etc. Subjective feedback will be collected in a questionnaire.

Instead of collecting subjective feedback in paper form the questions can be presented on a SmartPhone (Motorola Moto G) screen for those participants able to use a SmartPhone (Motorola Moto G). In that way the participant can answer the questions when he finds himself in a certain listening situation. Such a solution might be more comfortable than a paper questionnaire for some participants. An App for a mobile questionnaire called MobEval already exists from Phonak and will be used in this study. Participants will receive loaner SmartPhones (Motorola Moto G).

ELIGIBILITY:
Inclusion Criteria:

* all participants, which signed the Informed Consent (Appendix Informed Consent Form)
* severe to profound hearing impairment - bilaterally implanted with either the CII or HiRes90k cochlear implant devices
* experience with their more recent CI at least three months
* usage of the Naida CI sound processor on each ear for at least three months
* ability for speech understanding in the presence of competing noise without any assistance from lip-reading
* score: at least 20% correct for a sentence test delivered with an SNR of +10 dB, or an SRT of better (lower) than +15 dB
* ability to give subjective feedback in a certain listening situation
* first language: German or Swiss-German
* if participants are recruited additionally from other clinics, ability to travel to Zurich

Exclusion Criteria:

* Acute inflammation or pain in head-/neck area
* Dizziness
* Age of participants <18 years
* Age of participants > 80 years
* Any participant who is found to require substantial changes to their standard clinical program may be either excluded, or be asked to first get used to the new program before returning for the study test session.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: See below
Sampling Method: Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2016-10-31 (Actual); Study Completion 2016-10-31 (Actual)

PRIMARY OUTCOMES:
speech reception thresholds (SRT) assessment with audiological measures (omni) | 10 months
  The primary study outcome are speech reception thresholds (SRT) measured with omni-directional microphone setting
speech reception thresholds (SRT) assessment with audiological measures (BBF) | 10 months
  The primary study outcome are speech reception thresholds (SRT) measured with BBF microphone setting
speech reception thresholds (SRT) assessment with audiological measures (MBF) | 10 months
  The primary study outcome are speech reception thresholds (SRT) measured with MBF microphone setting

SECONDARY OUTCOMES:
paired comparisons assessment with scaling (speech intelligibility) | 10 months
  The main secondary outcome are paired comparisons which will be performed in the lab and on a guided tour outside the lab. The comparisons will be made with regards to speech intelligibility.
paired comparisons assessment with scaling (noise suppression) | 10 months
  The main secondary outcome are paired comparisons which will be performed in the lab and on a guided tour outside the lab. The comparisons will be made with regards to noise suppression.
paired comparisons assessment with scaling (overall) | 10 months
  The main secondary outcome are paired comparisons which will be performed in the lab and on a guided tour outside the lab. The comparisons will be made with regards to overall preference in each situation.

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Dillier, Prof. Dr, Principal Investigator — Universitätsspital Zürich, Klinik für ORL
Locations (1):
- Universitätsspital Zürich, Klinik für ORL, Zurich, Switzerland

REFERENCES:
- [Result] Buechner A, Dyballa KH, Hehrmann P, Fredelake S, Lenarz T. Advanced beamformers for cochlear implant users: acute measurement of speech perception in challenging listening conditions. PLoS One. 2014 Apr 22;9(4):e95542. doi: 10.1371/journal.pone.0095542. eCollection 2014. PMID 24755864
- [Result] Chung K, Zeng FG, Acker KN. Effects of directional microphone and adaptive multichannel noise reduction algorithm on cochlear implant performance. J Acoust Soc Am. 2006 Oct;120(4):2216-27. doi: 10.1121/1.2258500. PMID 17069317
- [Result] Chung K, Zeng FG. Using hearing aid adaptive directional microphones to enhance cochlear implant performance. Hear Res. 2009 Apr;250(1-2):27-37. doi: 10.1016/j.heares.2009.01.005. Epub 2009 Jan 22. PMID 19450437
- [Result] Chung K, Nelson L, Teske M. Noise reduction technologies implemented in head-worn preprocessors for improving cochlear implant performance in reverberant noise fields. Hear Res. 2012 Sep;291(1-2):41-51. doi: 10.1016/j.heares.2012.06.003. Epub 2012 Jun 28. PMID 22750449
- [Result] Compton-Conley CL, Neuman AC, Killion MC, Levitt H. Performance of directional microphones for hearing aids: real-world versus simulation. J Am Acad Audiol. 2004 Jun;15(6):440-55. doi: 10.3766/jaaa.15.6.5. PMID 15341225
- [Result] Kokkinakis K, Loizou PC. Multi-microphone adaptive noise reduction strategies for coordinated stimulation in bilateral cochlear implant devices. J Acoust Soc Am. 2010 May;127(5):3136-44. doi: 10.1121/1.3372727. PMID 21117762
- [Result] van der Beek FB, Soede W, Frijns JH. Evaluation of the benefit for cochlear implantees of two assistive directional microphone systems in an artificial diffuse noise situation. Ear Hear. 2007 Feb;28(1):99-110. doi: 10.1097/AUD.0b013e31802d0a55. PMID 17204902